CLINICAL TRIAL: NCT06697145
Title: Assessment of the Durability and Clinical Effectiveness of Parasympathetic Denervation Following Cardioneuroablation Using Physiological Indices of Heart Rate Reactivity
Brief Title: Assessment of the Durability of Cardioneuroablation Using Physiological Indices of Heart Rate Reactivity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wroclaw Medical University (Other)
Responsible Party: Principal Investigator, Piotr Niewinski, MD, MD, PhD, Wroclaw Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KB-331/2022
Record Dates: First submitted 2024-11-17; First posted 2024-11-20 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Syncope, Vasovagal, Neurally-Mediated
MeSH Terms: conditions — Syncope, Vasovagal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Cardioneuroablation (Experimental)
  Interventions: Procedure: Cardioneuroablation

INTERVENTIONS:
Procedure: Cardioneuroablation — Ablation of parasympathetic ganglia of the heart

SUMMARY:
Cardioneuroablation is a novel treatment option for reflex-mediated syncope. It involves thermal destruction of neural tissue in the close proximity of heart using catheter introduced to the heart through vein in the groin. Effectiveness of the procedure is satisfactory, however, in some cases there is a possibility of the re-growth of previously ablated tissue. We aim to investigate whether this process could be traced by measurement of various physiological parameters related to heart rate reactivity. Additionally we intend to reveal whether changes in those parameters over time could influence clinical effeciveness of the procedure.

ELIGIBILITY:
Inclusion Criteria:

* signed informed consent
* sinus rhythm
* clinical indications for cardioneuroablation for the treatment of vagally-mediated syncope

Exclusion Criteria:

* pregnancy
* known atropine hypersensitivity

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2021-11-23 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Change in degree of parasympathetic denervation (%) | 12 months

SECONDARY OUTCOMES:
Change in heart rate (beats/min) | 12 months
Change in heart rate variability (ms) | 12 months
Change in cardiac barosensitivity (ms/mmHg) | 12 months
Change in hypoxic heart rate response (beats/min SpO2) | 12 months
Time to recurrence of syncopal event (days | 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- Wroclaw Medical University, Wroclaw, Lower Silesian Voivodeship, Poland

IPD SHARING:
Plan to Share IPD: Undecided